CLINICAL TRIAL: NCT06917846
Title: Is Medical Therapy Alone Efficient for the Management of Medication-Related Osteonecrosis of the Jaw Bones (MRONJ) in All Stages?: A Comparative Study
Brief Title: Medical and Surgical Treatment of MRONJ (Medication-related Osteonecrosis of the Jaw Bones)
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alper Sindel, Professor, Akdeniz University
Other Study IDs: 2023/ KAEK-268
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Osteonecrosis Due to Drugs, Jaw; Osteonecrosis of the Jaw, Bisphosphonate Related; Osteonecrosis of the Jaw, Bisphosphonate Induced
Keywords: Antibiotics; Bisphosphonate; BRONJ; MRONJ; Osteonecrosis
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical treatment group: Sixty patients in this group were treated with antibiotherapy following oral hygiene instructions, which included daily chlorhexidine mouthwash recommendation in addition to routine oral hygiene measures.
  The systemic antibiotherapy spanned 3 weeks. Once the intraoral infection was contained and brought under control, the borders of the necrotic bone were expected to become more prominent and spontaneous sequestration was expected to follow. During follow-up controls, pus formation, pain status, lesion size, presence of spontaneous sequestration and recurrence were evaluated and recorded.
- Surgical treatment group: Forty-two patients were treated surgically. During follow-up controls, pus formation, pain status, lesion size, presence of spontaneous sequestration and recurrence were evaluated and recorded.

SUMMARY:
MRONJ is an acronym used to describe medication-related osteonecrosis of the jaw bones. It has been reported by the AAOMS that bisphosphonates or denosumab can cause this condition. The management of medication-related osteonecrosis of the jaw (MRONJ) is challenging, and there is ongoing debate over whether medical or surgical treatment is the gold standard. The aim of this retrospective study is to investigate the efficacies of medical and surgical treatments of MRONJ and comparatively evaluate their outcomes.

DETAILED DESCRIPTION:
This study analyzed 116 MRONJ lesions in 102 patients, divided into medical and surgical treatment groups. Sixty patients in medical treatment group were treated with antibiotherapy following oral hygiene instructions, which included daily chlorhexidine mouthwash recommendation in addition to routine oral hygiene measures.The systemic antibiotherapy spanned 3 weeks. Once the intraoral infection was contained and brought under control, the borders of the necrotic bone were expected to become more prominent and spontaneous sequestration was expected to follow. Forty-two patients were treated surgically. During follow-up controls, pus formation, pain status, lesion size, presence of spontaneous sequestration and recurrence were evaluated and recorded. Outcomes after 12 months were categorized into four healing response groups. (H1) Complete healing: Complete healing with a total coverage of previously exposed bone by the oral mucosa, (H2) Partial healing: Healthy progress for clinical outcomes and downstaging of the lesion according to the AAOMS criteria, (H3) Stable disease: No clinical alterations without any change for the clinical stage of the lesion, (H4) Progressive disease: Deteriorated clinical outcomes following lesion upstaging.

Associations between variables and outcomes were assessed using Chi-Square and Fisher's exact tests.

ELIGIBILITY:
Inclusion Criteria:

* Use of antiresorptive and/or antiangiogenic drugs and consequent development of MRONJ.
* Absence of head and neck radiotherapy.
* Presence of necrotic bone in the maxillofacial region for at least 8 weeks.

Exclusion Criteria:

* Having undergone head and neck radiotherapy.
* Presence of active radiotherapy and/or chemotherapy.
* Missing information in treatment and follow-up records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included 116 MRONJ lesions of different stages in 102 patients, who were referred to Akdeniz University, School of Dentistry, Department of Oral and Maxillofacial Surgery between January 2018 and January 2023. All patients had undergone anti-resorptive and/or anti-angiogenic drug treatment for various systemic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Healing status of MRONJ lesions after medical vs surgical treatment | Treatment outcomes were assessed after 12 months.
  To evaluate the effectiveness of medical versus surgical treatment in MRONJ patients by assessing the degree of healing (H1-H4) achieved after treatment.
  H1: Complete healing H2: Partial healing H3: Stabilization (Stagnation of the disease) H4: Progression (Disease progression)

SECONDARY OUTCOMES:
Correlation between spontaneous sequestration and healing | Treatment outcomes were assessed after 12 months.
  Spontaneous sequestration of osteonecrotic bone is expected in medically treated patients. Measurement of correlation between spontaneous sequestration and healing outcomes in medically treated MRONJ lesions.
Impact of MRONJ stage on treatment outcomes | Treatment outcomes were assessed after 12 months.
  The impact of MRONJ stage on treatment outcomes, specifically comparing the effectiveness of medical and surgical approaches in different disease stages.
Incidence of secondary osteonecrosis | Treatment outcomes were assessed after 12 months.
  Determination of the incidence of secondary osteonecrosis after surgical treatment, especially in stage 3 MRONJ lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Varoni EM, Lombardi N, Villa G, Pispero A, Sardella A, Lodi G. Conservative Management of Medication-Related Osteonecrosis of the Jaws (MRONJ): A Retrospective Cohort Study. Antibiotics (Basel). 2021 Feb 17;10(2):195. doi: 10.3390/antibiotics10020195. PMID 33671429
- [Background] Khan AA, Morrison A, Hanley DA, Felsenberg D, McCauley LK, O'Ryan F, Reid IR, Ruggiero SL, Taguchi A, Tetradis S, Watts NB, Brandi ML, Peters E, Guise T, Eastell R, Cheung AM, Morin SN, Masri B, Cooper C, Morgan SL, Obermayer-Pietsch B, Langdahl BL, Al Dabagh R, Davison KS, Kendler DL, Sandor GK, Josse RG, Bhandari M, El Rabbany M, Pierroz DD, Sulimani R, Saunders DP, Brown JP, Compston J; International Task Force on Osteonecrosis of the Jaw. Diagnosis and management of osteonecrosis of the jaw: a systematic review and international consensus. J Bone Miner Res. 2015 Jan;30(1):3-23. doi: 10.1002/jbmr.2405. PMID 25414052
- [Background] Junquera L, Gallego L, Cuesta P, Pelaz A, de Vicente JC. Clinical experiences with bisphosphonate-associated osteonecrosis of the jaws: analysis of 21 cases. Am J Otolaryngol. 2009 Nov-Dec;30(6):390-5. doi: 10.1016/j.amjoto.2008.07.014. Epub 2009 Mar 9. PMID 19880027
- [Background] Mucke T, Jung M, Koerdt S, Mitchell DA, Loeffelbein D, Kesting MR. Free flap reconstruction for patients with bisphosphonate related osteonecrosis of the jaws after mandibulectomy. J Craniomaxillofac Surg. 2016 Feb;44(2):142-7. doi: 10.1016/j.jcms.2015.11.015. Epub 2015 Dec 8. PMID 26752221
- [Background] Wilde F, Heufelder M, Winter K, Hendricks J, Frerich B, Schramm A, Hemprich A. The role of surgical therapy in the management of intravenous bisphosphonates-related osteonecrosis of the jaw. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Feb;111(2):153-63. doi: 10.1016/j.tripleo.2010.04.015. Epub 2010 Jul 31. PMID 20674411
- [Background] Vanpoecke J, Verstraete L, Smeets M, Ferri J, Nicot R, Politis C. Medication-related osteonecrosis of the jaw (MRONJ) stage III: Conservative and conservative surgical approaches versus an aggressive surgical intervention: A systematic review. J Craniomaxillofac Surg. 2020 Apr;48(4):435-443. doi: 10.1016/j.jcms.2020.02.017. Epub 2020 Mar 3. No abstract available. PMID 32178949
- [Background] Zirk M, Kreppel M, Buller J, Pristup J, Peters F, Dreiseidler T, Zinser M, Zoller JE. The impact of surgical intervention and antibiotics on MRONJ stage II and III - Retrospective study. J Craniomaxillofac Surg. 2017 Aug;45(8):1183-1189. doi: 10.1016/j.jcms.2017.05.027. Epub 2017 Jun 4. PMID 28684074
- [Background] Voss PJ, Joshi Oshero J, Kovalova-Muller A, Veigel Merino EA, Sauerbier S, Al-Jamali J, Lemound J, Metzger MC, Schmelzeisen R. Surgical treatment of bisphosphonate-associated osteonecrosis of the jaw: technical report and follow up of 21 patients. J Craniomaxillofac Surg. 2012 Dec;40(8):719-25. doi: 10.1016/j.jcms.2012.01.005. Epub 2012 Feb 14. PMID 22336489
- [Background] Hayashida S, Soutome S, Yanamoto S, Fujita S, Hasegawa T, Komori T, Kojima Y, Miyamoto H, Shibuya Y, Ueda N, Kirita T, Nakahara H, Shinohara M, Umeda M. Evaluation of the Treatment Strategies for Medication-Related Osteonecrosis of the Jaws (MRONJ) and the Factors Affecting Treatment Outcome: A Multicenter Retrospective Study with Propensity Score Matching Analysis. J Bone Miner Res. 2017 Oct;32(10):2022-2029. doi: 10.1002/jbmr.3191. Epub 2017 Jul 11. PMID 28585700
- [Background] Moretti F, Pelliccioni GA, Montebugnoli L, Marchetti C. A prospective clinical trial for assessing the efficacy of a minimally invasive protocol in patients with bisphosphonate-associated osteonecrosis of the jaws. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Dec;112(6):777-82. doi: 10.1016/j.tripleo.2011.07.004. Epub 2011 Oct 14. PMID 22000426
- [Background] Rodriguez-Lozano FJ, Onate-Sanchez RE. Treatment of osteonecrosis of the jaw related to bisphosphonates and other antiresorptive agents. Med Oral Patol Oral Cir Bucal. 2016 Sep 1;21(5):e595-600. doi: 10.4317/medoral.20980. PMID 27475683
- [Background] Carlson ER, Schlott BJ. Anti-resorptive osteonecrosis of the jaws: facts forgotten, questions answered, lessons learned. Oral Maxillofac Surg Clin North Am. 2014 May;26(2):171-91. doi: 10.1016/j.coms.2014.01.005. Epub 2014 Mar 13. PMID 24630868
- [Background] Ozalp O, Toru HS, Altay MA, Sindel A. Evaluation of the Efficacy of EDTA Chelation on Alveolar Bone Healing After Ultrasonic and Conventional Surgery Under Bisphosphonate Medication: A Rat Model. J Oral Maxillofac Surg. 2019 Oct;77(10):1982-1989. doi: 10.1016/j.joms.2019.04.011. Epub 2019 Apr 18. PMID 31095928
- [Background] Nicolatou-Galitis O, Schiodt M, Mendes RA, Ripamonti C, Hope S, Drudge-Coates L, Niepel D, Van den Wyngaert T. Medication-related osteonecrosis of the jaw: definition and best practice for prevention, diagnosis, and treatment. Oral Surg Oral Med Oral Pathol Oral Radiol. 2019 Feb;127(2):117-135. doi: 10.1016/j.oooo.2018.09.008. Epub 2018 Oct 9. PMID 30393090
- [Background] Ruggiero SL, Dodson TB, Aghaloo T, Carlson ER, Ward BB, Kademani D. American Association of Oral and Maxillofacial Surgeons' Position Paper on Medication-Related Osteonecrosis of the Jaws-2022 Update. J Oral Maxillofac Surg. 2022 May;80(5):920-943. doi: 10.1016/j.joms.2022.02.008. Epub 2022 Feb 21. PMID 35300956